CLINICAL TRIAL: NCT02362620
Title: Prospective Multi-centre Study of Prognostic Factors in Metastatic Castration-Resistant Prostate Cancer Patients Treated With Docetaxel or Cabazitaxel.
Brief Title: PROSTAC: Prospective Multi-centre Study of Prognostic Factors in mCRPC Patients Treated With Docetaxel or Cabazitaxel.
Acronym: PROSTAC
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Centro Nacional de Investigaciones Oncologicas CARLOS III (Other)
Responsible Party: Sponsor
Other Study IDs: CNI-DOC-2014-02; CNIO-CP-02-2014 (Other: CNIO)
Record Dates: First submitted 2015-02-09; First posted 2015-02-13 (Estimated); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Advanced Prostate Cancer; Cabazitaxel; Docetaxel
Keywords: metastatic Castration Resistant Prostate Cancer; Taxanes; Biomarkers

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood and FFPE tissue
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Docetaxel: Docetaxel 75mg/m2 IV every 3 weeks
- Cabazitaxel: Cabazitaxel 20-25mg/m2 IV every 3 weeks

SUMMARY:
PROSTAC is a prospective multicentre observational study in metastatic Castration-Resistant Prostate Cancer (mCRPC), designed to explore prognostic biomarkers in patients undergoing treatment with docetaxel or cabazitaxel

DETAILED DESCRIPTION:
This study is a prospective biomarker study of patients with mCRPC undergoing treatment with docetaxel or cabazitaxel as standard of care treatment. The participants will undergo serial pre- and post-therapy blood collection for biomarker analysis as part of the primary objective of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Male age ≥ 18 years
2. Histologically confirmed adenocarcinome of the prostate
3. ECOG Performance Status ≤ 2
4. Castration resistance must be documented with surgical or medical castration with serum testosterone < 50 ng/mL (< 2.0 nM).
5. Men diagnosed with at least one metastatic lesion on CT or bone scan.
6. Documented biochemical and/or radiographic progression to previous treatment according to PCWG2 criteria.
7. Patients who are candidates for standard of care treatment with docetaxel 75mg/m2 every 3 weeks or cabazitaxel 20-25mg/m2 every 3 weeks intravenously.
8. Availability of formalin-fixed paraffin-embedded blocks from the prostate biopsy and/or radical prostatectomy.
9. Acceptable hematological, hepatic and renal functions.

Exclusion Criteria:

1. Previous cancer diagnosis, except those patients who had a localized malignant tumour and who are five years cancer-free or those diagnosed with skin cancers (of non-melanoma type) or excised in situ carcinomas.
2. Any condition or reason that, in the opinion of the Investigator, interferes with the ability of the patient to participate in the trial, which places the patient at undue risk, or complicates the interpretation of safety data

Ages: 18 Years to 99 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Castration-Resistant Prostate Cancer patients
Sampling Method: Non-Probability Sample
Enrollment: 402 (Estimated)
Dates: Start 2014-05; Primary Completion 2018-04 (Actual); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
To validate the prognostic value of the gene-expression signature from peripheral blood described by Olmos et al (Lancet Oncol 2012) on overall survival of mCRPC patients | 48 months

SECONDARY OUTCOMES:
To analyze the prognostic value of the gene-expression signature described by Olmos et al on biochemical and radiological progression-free survival | 48 months
To analyze the prognostic value of early changes in the gene-expression signature described by Olmos et al | 48 months
To compare the prognostic value of the gene-expression signature described by Olmos et al versus the gene-expression signature described by Ross et al (Lancet Oncol, 2012) | 48 months
To validate the prognostic value of classical nomograms designed to assess the outcomes of mCRPC patients in these both cohorts of patients | 48 months
To analyze the prognostic value of TMPRSS2-ERG rearrengement and PTEN loss in these cohorts | 48 months
To analyze the prognostic value of AR splicing variants, serum chromogranine and serum testosterone levels measured by ultrasensitive method in these both cohorts of patients | 48 months
To correlate the presence of somatic and/or germinal mutations with the outcomes of these patients | 48 months

CONTACTS AND LOCATIONS:
Overall Officials: David Olmos, MD, PhD, Principal Investigator — Head of Prostate Cancer Clinical Research Unit CNIO
Locations (25):
- Spain (25):
  - Hospital Universitario de Santiago, Santiago de Compostela, A Coruña
  - ICO L'Hospitalet, L'Hospitalet de Llobregat, Barcelona
  - Hospital Althaia Manresa, Manresa, Barcelona
  - Hospital de Especialidades de Jerez de la Frontera, Jerez de la Frontera, Cádiz
  - Hospital Costa del Sol, Marbella, Málaga
  - Complejo Hospitalario de Navarra, Pamplona, Navarre
  - Hospital Universitario de Canarias, San Cristóbal de La Laguna, Tenerife
  - Fundacion Centro Oncologico de Galicia, A Coruña
  - Hospital Universitario Vall D'Hebron, Barcelona
  - Hospital de Ciudad Real, Ciudad Real
  - Hospital Universitario Reina Sofia, Córdoba
  - Hospital Universitario Virgen de las Nieves, Granada
  - Hospital Universitario de Guadalajara, Guadalajara
  - Hospital Universitario Gregorio Maranon, Madrid
  - Coordination PROCURE-Centro Nacional de Investigaciones Oncologicas, Madrid
  - Hospital Universitario Clinico San Carlos, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Centro Integral Oncológico Clara Campal, Madrid
  - Anatomical Pathology PROCURE, Málaga
  - Hospital Regional Universitario Virgen de la Victoria, Málaga
  - Hospital Universitario Virgen de la Victoria, Málaga
  - Hospital Morales Messeguer, Murcia
  - Hospital Son Espases, Palma de Mallorca
  - Complejo Hospitalario de Pontevedra, Pontevedra
  - Hospital Universitario La Fe, Valencia